CLINICAL TRIAL: NCT03896100
Title: Assessment of Levels of Intracellular Cytokines and Markers in Cells Recovered From the Anterior Eye (Phase 3)
Brief Title: Assessment of Intracellular Cytokines and Markers in Cells (Phase 3)
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR-6315
Record Dates: First submitted 2019-03-28; First posted 2019-03-29 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Impression Cytology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — ocular surface cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Element 2: Four clinical samples will be taken from each eligible subject and used to assess two clinical removal methods and two in vitro removal methods.
- Element 3: Four clinical samples will be taken from each eligible subject and used to assess three different storage methods.
- Element 4: Four clinical samples will be taken from each eligible subject and used to assess different ocular regions.

SUMMARY:
This is a single arm, prospective, bilateral, non-randomized study that will be split into four elements. Element 1 will be an in vitro non-clinical study and described in the laboratory protocol. Elements 2, 3 and 4 will each be a single non-dispensing visit.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. They are of legal age (18 years) and capacity to volunteer.
  2. They understand their rights as a research subject and are willing and able to sign a Statement of Informed Consent.
  3. They are willing and able to follow the protocol.
  4. They agree not to participate in other clinical research for the duration of this study.

     Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. They have had cataract surgery.
  2. They have had corneal refractive surgery.
  3. They have any corneal distortion resulting from previous hard or rigid lens wear or have keratoconus.
  4. They are pregnant or breast-feeding.
  5. They have any infectious disease (e.g. hepatitis) or any immunosuppressive disease (e.g. HIV) or a history or anaphylaxis or severe allergic reactions.
  6. They have taken part in any other contact lens or care solution clinical trial research, within two weeks prior to starting this study.
  7. They are currently regularly (once per day or more) using oral or inhaled steroids or anti-inflammatory medications.
  8. They are using any topical medications such as eye drops or ointments.
  9. They are a current (i.e. within the last three months) contact lens wearer (wearing a lens in one or both eyes).
  10. History of allergic reaction to sodium fluorescein or topical anesthetic.
  11. They have Grade 3 or greater of any of the following ocular surface signs: corneal edema, corneal vascularization, corneal staining (white light evaluation), tarsal conjunctival changes or any other abnormality which would normally contraindicate contact lens wear.
  12. Any active ocular infection or inflammation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible subjects aged 18 years and above with normal healthy eyes will be recruited for this work.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Number of Cells | 1.5 hours duration of assessment time
  The frequency count of cells will be summarized within the category.
Types of Cells | 1.5 hours duration of assessment time
  The percentage of types of cells will be summarized within the category.

CONTACTS AND LOCATIONS:
Locations (1):
- Eurolens Research - The University of Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu